CLINICAL TRIAL: NCT07379619
Title: Improving Neonatal Transport Knowledge of Neonatal Intensive Care Unit Nurses and Physicians Using a Safe Transport Algorithm and Physiological Stability Transport Risk Index: A Quasi-experimental Study
Brief Title: Safe Transport Algorithm and TRIPS in Neonatal Transport
Acronym: TRIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beste Ozguven Oztornaci (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Sponsor-Investigator, Beste Ozguven Oztornaci, Assist. Prof. Dr., Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22.09.2022/0379
Record Dates: First submitted 2026-01-11; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Nursing; Transportation of Patients; Newborn
Keywords: Pediatric Nursing; Newborn; Transportation; Knowledge

STUDY DESIGN:
Intervention Model Description: Quasi-experimental (single-group pretest-posttest) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- involving a total of 100 volunteer healthcare professionals, including 72 nurses and 28 physicians (Experimental): Pre-intervention, data were collected in two stages, before and after training, using a 33-item "Newborn Transport Knowledge Assessment Form" developed by researchers and validated based on expert opinions. As part of the intervention, a 10-step safe transport algorithm developed by researchers and validated by expert opinion, along with TRIPS, was displayed in clinical areas, and verbal training was provided to participants. Post intervention, data were collected in two stages, before and after training, using a 33-item "Newborn Transport Knowledge Assessment Form".
  Interventions: Behavioral: As part of the intervention, a 10-step safe transport algorithm developed by researchers and validated by expert opinion, along with TRIPS, was displayed in clinical areas, and verbal training was pro

INTERVENTIONS:
Behavioral: As part of the intervention, a 10-step safe transport algorithm developed by researchers and validated by expert opinion, along with TRIPS, was displayed in clinical areas, and verbal training was pro — In this intervention, a 10-step safe transport algorithm developed by researchers and approved by expert opinion was used. In addition, the TRIPS index, which was not used as standard practice at the clinic where the research was conducted, began to be used as part of the intervention.

SUMMARY:
Aim: Newborn babies may need to be referred to different centers to receive the care they need. It is important to improve the quality of neonatal transport to reduce infant mortality rates. This study was conducted to examine the effect of the use of transport algorithm and TRIPS (Transport Risk Index of Physiological Stability) on the knowledge level of nurses and physicians working in the neonatal intensive care unit.

DETAILED DESCRIPTION:
The following hypotheses were tested within the scope of the research:

H1: Using structured educational interventions that include the "Safe Transport Algorithm" increases the knowledge level of neonatal nurses and physicians regarding neonatal transport.

H2: Using structured educational interventions that include the "Transport Physiological Stability Risk Index (TRIPS)" increases the knowledge level of neonatal nurses and physicians regarding neonatal transport.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate voluntarly in the study and working as a nurse or physician in the neonatal intensive care unit.

Exclusion Criteria:

* Change in the participant's workplace during the data collection process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Knowledge Level Assessment Form on Neonatal Transport Form | 1 month
  This form has been developed by researchers in line with the relevant literatüre. The form consists of a total of 33 items aimed at assessing the level of knowledge regarding newborn transport. Participants were asked to select one of the options "true," "false," or "I don't know" for each item. Correct answers are worth 1 point, while incorrect answers and "I don't know" responses are worth 0 points. The total possible score on the form ranges from 0 to 33. In order to evaluate the validity of the forms, the final version of the forms was determined by consulting experts. The minimum Coverage Validity Ratio (CVR) is accepted as 0.99. The 19 items with low CVR values were revised and resubmitted to the experts for approval. As a result of the final evaluation, the Content Validity Index calculated based on the CVR average of the items was found to be 1.00, and it was determined that the content validity of the form was statistically sufficient.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Izmir, ÇİĞLİ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No